CLINICAL TRIAL: NCT04204915
Title: A Randomised Controlled Trial of Early Valve Replacement in Severe ASYmptomatic Aortic Stenosis
Brief Title: The Early Valve Replacement in Severe ASYmptomatic Aortic Stenosis Study
Acronym: EASY-AS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University of Auckland, New Zealand (Other); University Hospitals, Leicester (Other); The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0700; CS/18/7/33714 (Other Grant/Funding Number: British Heart Foundation); 266292 (Other: IRAS); 90865 (Other: EDGE); 0700 (Other: Sponsor)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis
Keywords: Asymptomatic aortic stenosis; Aortic valve replacement; Randomised controlled trial; Expectant management; Hospitalisation for heart failure; Cardiovascular death
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Aortic valve replacement (Active Comparator): Participants randomised to AVR will be investigated and managed according to local protocols and standard practice. Participants will be placed on the waiting list with the aim that surgery will be performed within 3 months, dependent on local hospitals' waiting lists.
  Interventions: Procedure: Aortic valve replacement
- Group B: Expectant management (No Intervention): Participants randomised to expectant management will continue to have regular monitoring of their condition in line with the procedures and standard practices of their hospital.

INTERVENTIONS:
Procedure: Aortic valve replacement — Participants will be assessed by a member of the surgical team performing aortic valve replacement (AVR), and by any other relevant medical professionals identified by the doctors overseeing their care in hospital. When deemed ready for AVR, a member of the surgical team will ask for consent to proceed with the AVR. They will discuss the surgical procedure, covering information on the basic technical procedure, risks and expected recovery time.
  Arms: Group A: Aortic valve replacement

SUMMARY:
Aortic stenosis (AS) affects approximately 5% of individuals >65 years old, with ~3% of people >75 years having moderate to severe disease. The prevalence of AS is rising rapidly due to an ageing population and is projected to double in the next two decades. Increasingly clinicians face the dilemma of how to best manage this growing population of mainly elderly patients, many of whom are asymptomatic but have been identified as having severe AS, often as an incidental finding. Reduced aortic valve opening progresses over decades without any apparent symptoms because the heart compensates for the AS. Ultimately, compensatory mechanisms fail resulting in angina, syncope or heart failure. If these symptomatic patients with severe AS remain untreated, they have a dire prognosis. In this situation the only effective treatment is AVR, either surgically or using TAVI. Conversely, conventional teaching and clinical practice in cardiology has been that, in the absence of symptoms, the prognosis is usually excellent and, except in a few very specific circumstances, conservative management and regular review (expectant management) is recommended. This advice is reflected in current international guidelines but is based largely on historical precedent. There has never been a randomised controlled trial to address the relative benefits of early AVR versus expectant management in patients with severe asymptomatic AS. The relative benefits of a strategy of early AVR/TAVI versus expectant management in patients with asymptomatic severe AS are unclear. There is clinical equipoise but it remains one of the few areas of cardiovascular medicine where no randomised controlled trials (RCT) have been performed. The EASY-AS study will provide crucial data on the relative merits of these differing approaches to management, in terms of important patient orientated outcomes, conventional cardiovascular end-points and cost effectiveness.

DETAILED DESCRIPTION:
This is a major pragmatic multi-centre prospective parallel group open RCT. It will be conducted in the UK, Australia and New Zealand, funding is being sought in several countries to expand recruitment internationally. The study is in 2 phases: the vanguard and main phase. Therefore the study will run an internal pilot to prove recruitment of the relevant number of participants during the initial 2 years.

The over-arching aim is to determine whether early AVR results in better clinical outcomes and cost-effectiveness than a strategy of expectant management in asymptomatic patients with severe AS.

The primary hypothesis is that early AVR or TAVI in asymptomatic patients with severe AS will result in a reduction in the composite primary outcome of cardiovascular (CV) death and hospitalisation for heart failure (HHF) when compared to the conventional approach of expectant management.

Potential participants will be identified by a member of the clinical care team following diagnosis with severe AS. Participants will be screened for eligibility using pre-specified inclusion/exclusion criteria. Eligible participants will be provided with a written version of the participant information sheet detailing the exact nature of the study, what it will involve for the participant and any risks involved with taking part. Participants will be given at least 24 hours to consider the information and decide whether or not to take part. The study will randomise up to 2844 patients with severe asymptomatic AS to either allocated expectant management OR aortic valve replacement. Participants randomised to AVR will be placed on a waiting list with the aim that surgery will be performed within 3 months, dependent on local hospitals' waiting lists. Participants randomised to AVR will undergo routine tests/procedures which may include coronary angiography. If the outcome of the coronary angiography reveals coronary heart disease, the decision to perform CABG or PCI will be made by the responsible cardiac surgeon and cardiologist, in consultation with the patient. All analyses will be undertaken using the principles of intention-to-treat with participants analysed in the group they were randomised regardless of treatment received.

EASY-AS is collaborating with the EVoLVeD study (Early Valve Replacement guided by Biomarkers of Left Ventricular Decompensation in Asymptomatic Patients with Severe Aortic Stenosis, Clinical Trials.gov NCT03094143). In centres where both EASY-AS and EVoLVeD are running, participants in EASY-AS will be offered the opportunity to take part in EVoLVeD.

Funding has been granted by the British Heart Foundation (UK), Medical Research Future Fund (Aus) and Heart Foundation (NZ). The UK sponsor is the University of Leicester. Additional support and resources for the study will be provided by the participating Trusts and their corresponding Clinical Research Networks in the UK. The central co-ordination centre is the University of Leicester Clinical Trials Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patient has severe asymptomatic AS, in line with current international guidelines, defined as either:

   1. Peak velocity ≥4m/s OR mean pressure gradient ≥40mmHg WITH aortic valve area ≤1.0cm2 OR ≤0.6cm2/m2 body surface area OR
   2. Peak velocity ≥4m/s OR mean pressure gradient ≥40mmHg WITH aortic valve area >1.0 - ≤1.2cm2 OR >0.6 - ≤0.7cm2/m2 body surface area AND high sex specific calcium score* OR
   3. Peak Velocity ≥3.5m/s - 3.9m/s AND mean pressure gradient <40 mmHg WITH aortic valve area ≤1.0cm2 OR ≤0.6cm2/m2 body surface area AND high sex specific calcium score* *Sex specific high calcium scores (Agatston units): >1200 females; >2000 males
3. The responsible clinician feels that either ongoing surveillance or early AVR are appropriate.
4. Regarded by the treating cardiologist to be suitable for AVR (surgical or TAVI) with an acceptable risk
5. Willing to provide informed consent and be randomised to early AVR or expectant management
6. An ability to understand one of the written languages that the study has provided written and visual materials in, or the availability of a translator to explain the study documentation

   Exclusion Criteria:
7. Symptoms related to AS
8. Additional severe valvular heart disease
9. Other cardiac surgery planned pre-randomisation (eg CABG)
10. Left ventricular systolic dysfunction (LVEF <50%)
11. Pregnancy
12. Co-morbid condition that, in the opinion of the treating cardiologist, limits life expectancy to <2 years
13. Patient has previously undergone AVR or TAVI with restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2844 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2031-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Combined measure of cardiovascular death and hospitalisation for heart failure | Minimum 3 years
  Measured in days from randomisation until end of trial (minimum 3 years).
  The primary analysis will be undertaken when 663 events have accrued, which is estimated to be after a median of 5 years follow-up assuming 2844 patients are recruited over 4 years.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS 2.0) | 6, 12, 24 and 36 months
  Assessing disability-free survival during the period of active recruitment.
  Scores assigned to each of the items - "none" (0), "mild" (1) "moderate" (2), "severe" (3) and "extreme" (4) - are summed. The simple sum of the scores of the items across all domains constitutes a statistic that is sufficient to describe the degree of functional limitations.
  Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
NHS record linkage services | Up to 5 years
  Assessing number of days alive and out of hospital.
  All participants will be consented for long-term follow-up (10 years) and clinical events will be ascertained through NHS Digital or equivalent.
Death (cardiovascular, including sudden cardiac death, and non-cardiovascular), hospitalisation for heart failure, myocardial infarction, stroke | Up to 5 years
  Assessing number of major adverse events.
  All participants will be consented for long-term follow-up (10 years) and clinical events will be ascertained through NHS Digital or equivalent.
Number of additional outcomes of special interest: infective endocarditis and major bleeding, resuscitated cardiac arrest, hospitalisation with new onset atrial fibrillation, syncope, revascularization (CABG/PCI), cardiac device implantation | Up to 5 years
  Assessing additional outcomes of special interest.
  All participants will be consented for long-term follow-up (10 years) and clinical events will be ascertained through NHS Digital or equivalent.
EuroQol five-level (EQ-5D-5L) questionnaire | 6, 12, 24 and 36 months
  Assessing quality of life during the period of active recruitment.
  EQ-5D-5L has 2 components: health state description and evaluation. In the description part, health status is measured in terms of 5 dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a 5-level scale.
Health Economics Questionnaire | 6, 12, 24 and 36 months
  Assessed using self-reported health care resource use and cost effectiveness.
  Participants will be asked if they have used any of the following services at a hospital for reasons that may be related to their heart condition or treatment: hospital services, services in the community and specialist equipment.
  The data from this questionnaire will be scored by a Health Economist at the end of the study.
Edmonton Frail Scale (EFS) (Bedside and Acute Care Version) | Baseline
  Assessing frailty at baseline using a simple tool to assess frailty in older patients. It consists of nine domains and eleven items, each scoring 0 points (frailty absent or normal health), 1 point (minor errors or mild/moderate impairment), or 2 points (important errors or severely impaired).

CONTACTS AND LOCATIONS:
Overall Officials: Gerry McCann, Prof, Principal Investigator — University of Leicester; Graham Hillis, Prof, Principal Investigator — The University of Western Australia; Ralph Stewart, Prof, Principal Investigator — University of Aukland
Locations (110):
- Australia (20):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Townsville Hospital, Douglas, Queensland
  - The Gold Coast Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Lyell McEwin Hospital, Elizabeth Vale
  - Northern Hospital, Epping
  - Royal Hobart Hospital, Hobart
  - Nepean Hospital, Kingswood
  - John Hunter Hospital, New Lambton Heights
  - Royal Darwin Hospital, Tiwi
- Belgium (3):
  - Sint-Jan Hospital, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospital of Brussels, Jette
- Netherlands (2):
  - Frisius Medical Center, Leeuwarden
  - Radboud University Medical Center, Nijmegen
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- Institute of Cardiovascular Diseases, Kamenitz, Serbia
- Spain (2):
  - Hospital Germans Trias, Barcelona
  - University Hospital of Navarra, Pamplona
- United Kingdom (79):
  - University Hospital of North Durham, Durham, County Durham
  - Glan Clwyd Hospital, Bodelwyddan, Denbighshire
  - Dorset County Hospital, Dorchester, Dorset
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - University Hospitals Leicester, Glenfield, Leicester, Leicestershire
  - Royal Liverpool Hospital, Liverpool, Merseyside
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Scunthorpe General Hospital, Scunthorpe, North Lincolnshire
  - Kettering General Hospital, Kettering, Northamptonshire
  - Wansbeck General Hospital, Ashington, Northumberland
  - Raigmore Hospital, Inverness, Scotland
  - Musgrove Park Hospital, Taunton, Somerset
  - Morriston Hospital, Swansea, Wales
  - Russells Hall Hospital, Dudley, West Midlands
  - George Eliot Hospital, Nuneaton, West Midlands
  - Walsall Manor Hospital, Walsall, West Midlands
  - Sandwell General Hospital, West Bromwich, West Midlands
  - Wycombe Hospital, High Wycombe, Wycombe
  - Aberdeen Royal Infirmary, Aberdeen
  - Aintree University Hospital, Aintree
  - University Hospital Ayr, Ayr
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Basildon University Hospital, Basildon
  - Queen Elizabeth Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Royal Sussex County Hospital, Brighton
  - North Cumbria Integrated Care, Carlisle
  - Chesterfield Royal Hospital, Chesterfield
  - University Hospital Coventry & Warwickshire, Coventry
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - Doncaster Royal Infirmary, Doncaster
  - Ninewells Hospital, Dundee
  - The Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Gateshead Health NHS Foundation Trust, Gateshead
  - Golden Jubilee National Hospital, Glasgow
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Hospitals NHS Foundation, Gloucester
  - Huddersfield Royal Infirmary, Huddersfield
  - West Middlesex University Hospital, Isleworth
  - Airedale General Hospital, Keighley
  - University Hospital Crosshouse, Kilmarnock
  - Leeds General Infirmary, Leeds
  - Lincoln County Hospital, Lincoln
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Liverpool Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - St Thomas' Hospital, London
  - University Hospital Lewisham, London
  - Chelsea and Westminster Hospital, London
  - St George's Hospital, London
  - Cleveland Clinic London Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Maidstone & Tunbridge Wells Hospital, Maidstone
  - Wythenshawe Hospital, Manchester
  - North Manchester General Hospital, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Kings Mill Hospital, Nottingham
  - Queens Medical Centre, Nottingham
  - Royal Alexandra Hospital, Paisley
  - Derriford Hospital, Plymouth
  - Poole Hospital, Poole
  - Queen Alexandra Hospital, Portsmouth
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Forth Valley Royal Hospital, Stirling
  - Stepping Hill Hospital, Stockport
  - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland
  - Torbay Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Pinderfields Hospital, Wakefield
  - South Warwickshire University NHS Foundation Trust, Warwick
  - Watford General Hospital, Watford
  - New Cross Hospital, Wolverhampton
  - Worcester Acute Hospitals NHS FT, Worcester
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allmark P, Taylor B, Tod AM, Ryan T, Dweck M, McCann GP, Singh A. Factors influencing the decision to accept or decline aortic valve replacement for asymptomatic aortic stenosis: a nested longitudinal qualitative substudy of the EASY-AS randomised trial. BMJ Open. 2026 Jan 22;16(1):e106485. doi: 10.1136/bmjopen-2025-106485. PMID 41571417